CLINICAL TRIAL: NCT03303274
Title: A Difference in the Cross-section Area of Subclavian Vein Between Supine and Lateral Tilt Position: Its Clinical Impact on Subclavian Venous Catheterization - Stage II
Brief Title: A Difference in Subclavian Vein Catheterization Between Supine and Lateral Tilt Position - Stage II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1707-110-871-2
Record Dates: First submitted 2017-09-25; First posted 2017-10-06 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Catheterization; Posture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipsilateral tilt (Experimental): The operation table will be tilted 20 degrees right laterally before subclavian venous catheterization.
  Interventions: Procedure: Ipsilateral tilt
- Supine (No Intervention): Catheterization of right subclavian vein in supine position.

INTERVENTIONS:
Procedure: Ipsilateral tilt — The operation table will be tilted 20 degrees right laterally.
  Arms: Ipsilateral tilt

SUMMARY:
Central venous catheterization is widely used for various purposes during surgery. For central venous catheterization, subclavian vein is selected because of the relatively low risk of infection, long-term patency and low patient discomfort. The cross - sectional area of the subclavian vein is an important factor to increase success rate. Several studies have reported that the Trendelenburg position increases the cross-sectional area of the subclavian vein, and the lateral tilt position can change the cross-sectional area of the subclavian vein. However, the impact of lateral tilt position to the cross-sectional area of the subclavian vein is not clear. The ipsilateral position can increase the cross-sectional area of the subclavian vein, and the contralateral position can decrease the cross-sectional area by gravity.

In the second stage of this study, the investigators would like to compare the success rate, the number of needle passage, time to complete subclavian vein catheterization in supine and ipsilateral tile position.

ELIGIBILITY:
Inclusion Criteria:

- the patients who receive elective neurosurgical surgery and require central venous catheter

Exclusion Criteria:

* the patients who have puncture site infection
* the patients who have chemoport, pacemaker in right subclavian vein
* the patients who had received right mastectomy or right pneumonectomy
* other contraindications for subclavian venous catheterization (eg. mass, hematoma, vegetation, and anticoagulation)

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-10-20 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
The number of needle passage | during subclavian venous catheterization
  The number of needle passage for puncture of subclavian vein

SECONDARY OUTCOMES:
Time to puncture subclavian vein | during subclavian venous catheterization
  Time to puncture subclavian vein
Time to insert guidewire | during subclavian venous catheterization
  Time to insert guidewire
Time to insert dilator | during subclavian venous catheterization
  Time to insert dilator
The number of trial to insert catheter | during subclavian venous catheterization
  The number of trial to insert catheter
Time to insert catheter | during subclavian venous catheterization
  Time to insert catheter
Success of catheter insertion | during subclavian venous catheterization
  Final success of catheter insertion within 6 trials
Other complications with central venous catheterization | From subclavian venous catheterization to 24 hours after operation finished
  complications with central venous catheterization such as arterial puncture, perivascular hematoma, pneumothorax, and malpositioning

REFERENCES:
- [Derived] Yoon HK, Lee HC, Kang P, Lee JM, Park HP, Cho YJ. Effects of ipsilateral tilt position on the cross-sectional area of the subclavian vein and the clinical performance of subclavian vein catheterization: a prospective randomized trial. BMC Anesthesiol. 2020 Sep 5;20(1):226. doi: 10.1186/s12871-020-01144-1. PMID 32891115
- [Derived] Jung DE, Lee HC, Yoon HK, Park HP. The effects of ipsilateral tilt position on right subclavian venous catheterization: study protocol for a prospective randomized trial. Trials. 2018 May 24;19(1):292. doi: 10.1186/s13063-018-2666-8. PMID 29793550